CLINICAL TRIAL: NCT03645811
Title: Music Therapy and EFT: Integrative Medicine on Exam Anxiety in Turkish Nursing Students
Brief Title: Integrative Medicine on Exam Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Demet İnangil, PhD, Assistant Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 10840098-604.01.01-E.11892
Record Dates: First submitted 2018-08-09; First posted 2018-08-24 (Actual); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Educational Problems
Keywords: anxiety; OSCE; EFT; music
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Students who arrived on the day of the exam were assigned to the music therapy (M1 and M2), and EFT (E1 and E2) groups, and the control group (K1 and K2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Implementation of music therapy (Experimental): For the music therapy, lecturers specializing in music therapy were consulted and accordingly a "mahur maqam," an instrumental piece of traditional Turkish music played on the saz, was chosen. The mahur maqam has a descending scale, which has a relaxing impact as it moves along a 1-2 octave sound spectrum. It elicits feelings of joy and positivity, and immediately draws the attention of the listener, helping keep the mind clear. The mahur maqam belongs to the rast maqam family. Rast maqams are usually evocative of feelings of peacefulness, surrender, tranquility, trust, and mystical sentiments.
  Interventions: Behavioral: Music Therapy
- Implementation of EFT (Experimental): The EFT application protocol was explained to the students with the help of the image in the picture for 5 minutes. The method was applied through the investigator tapping on their bodies and the students repeating the steps for three sessions. Each of the treatment sessions was approximately three minutes, resulting in a nine-minute treatment for intervention. Each EFT session was performed by following the steps below.
  The content of each EFT session was as follows:
  1. Preparation
  2. Tapping Series
  3. The Nine Gamut Sequence and Eye Movements
  Interventions: Behavioral: EFT
- Control (No Intervention): For the control group, 15 minutes of free time was given.

INTERVENTIONS:
Behavioral: Music Therapy — Music therapy was applied in the application room. Via a portable computer, students listened to the mahur maqam for 20 minutes under the supervision of the investigators using an MP3 player.
  Arms: Implementation of music therapy
Behavioral: EFT — EFT includes taps, nine gamut sequences, and eye movements on the meridian system, focusing on the individual's inhibiting thoughts, disturbing emotions, or memories. EFT regulates the flow of energy in the meridian system of the individual, causing relaxation in the mind, body, and emotions.
  Arms: Implementation of EFT

SUMMARY:
Introduction: Test anxiety, one of the forms of situational anxiety, is a crucial biopsychological factor negatively affecting the wellbeing and academic performance of students throughout their education. The study aims to determine the effects of music therapy and EFT (Emotional Freedom Technique) on situational anxiety and vital signs in nursing students before they take the OSCE (Objective Structured Clinical Exam).

The study was a randomized controlled experimental study and conducted with 90 volunteering students studying at the Faculty of Health Sciences, Department of Nursing at a university in Istanbul. A computer-based random number generator was used to randomly assign the students into three groups (Music, EFT, and control), each of which consisted of 30 students. Data collection was carried out using a Student Identification Form, the Situational Anxiety Scale, and the Vital Signs Form.

DETAILED DESCRIPTION:
Anxiety - an important concept for describing human behaviors - is a condition in which a number of physiological responses are generated, accompanied by feelings of distress, anxiety, and depression in various scenarios where one feels threatened. Test anxiety experienced by nursing students around the world during their training is one of the most significant problems that hinder the acquisition of professional skills. Students in most nursing programs show poor exam performance due to anxiety caused by the OSCE exam. Studies on test anxiety also show a negative relationship between test anxiety and academic performance. When the literature is examined, it can be seen that stress reduction is very important in allowing students to maximize their learning of practical skills in the vocational education process. Techniques such as music therapy, cognitive therapy, emotional freedom technique (EFT), breathing techniques, mind cleansing, aromatherapy, and relaxation of muscles have been used to reduce the anxiety levels of nursing students . Based on prior research, the aim of the study to determine the effects of the music therapy and EFT (Emotional Freedom Technique), on situational anxiety and vital signs, before the OSCE (Objective Structured Clinical Exam) in nursing students.

This study was conducted with 90 volunteer students studying at the Nursing Department of the Health Sciences Faculty at a foundation university in Medipol University. The data was collected prior to the OSCE on May 31, 2017. Students included in the study were required to meet the eligibility criteria of (a) being 18 years old or above, (b) taking the theoretical course of Nursing Principles I and II, and (c) entering the OSCE on May 31 as part of the Nursing Principles course. All students taking the exam were included in the study without reverting to the method of sample size selection (n = 90). A randomly ordered class list was prepared with the student numbers in the classroom list using the random.org program. According to the newly created list, students were notified in writing one day before about what time to arrive before the exam. Students who arrived on the day of the exam were assigned to the music therapy and EFT groups, and the control group. Each group consisted of 30 students. The students were taken to a 90 m2 practice room. Each group was briefed for five minutes before obtaining their consent. The students had their vital signs measured by the investigators. They were asked to fill out the Student Identification Form and the Situational Anxiety Scale. Afterward, the methods (music and EFT) were applied for 15 minutes. The methods were applied by the investigators who are experts in their fields. After the methods were applied, the students had their vital signs remeasured by the investigators and were asked to fill out the Situational Anxiety Scale. For the control group, pre-measurements were taken, 15 minutes of free time was given, and then post-measurements were taken.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old or above,
* taking the theoretical course of Nursing Principles I and II,
* entering the OSCE on May 31 as part of the Nursing Principles course.

Exclusion Criteria:

* did not volunteer to participate in the study
* arrived late or did not turn up

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demet İnangil, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Medipol Universtiy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torabizadeh C, Bostani S, Yektatalab S. Comparison between the effects of muscle relaxation and support groups on the anxiety of nursing students: A randomized controlled trial. Complement Ther Clin Pract. 2016 Nov;25:106-113. doi: 10.1016/j.ctcp.2016.09.001. Epub 2016 Sep 7. PMID 27863599
- [Background] Ince S, Cevik K. The effect of music listening on the anxiety of nursing students during their first blood draw experience. Nurse Educ Today. 2017 May;52:10-14. doi: 10.1016/j.nedt.2017.02.009. Epub 2017 Feb 14. PMID 28214664
- [Background] Patterson SL. The effect of emotional freedom technique on stress and anxiety in nursing students: A pilot study. Nurse Educ Today. 2016 May;40:104-10. doi: 10.1016/j.nedt.2016.02.003. Epub 2016 Feb 7. PMID 27125158

RESULTS

PARTICIPANT FLOW:
Groups:
- Music Therapy: In the study, music therapy was applied in the application room. Via a portable computer, students listened to the mahur maqam for 15 minutes under the supervision of the investigators using an MP3 player.
  Music Therapy: Music therapy was applied in the application room. Via a portable computer, students listened to the mahur maqam for 20 minutes under the supervision of the investigators using an MP3 player.
- Emotional Freedom Technique: The EFT application protocol was explained to the students with the help of the image in the picture. The method was applied through the investigators tapping on their bodies and the students repeating the steps.
  EFT: EFT includes taps, nine gamut sequences, and eye movements on the meridian system, focusing on the individual's inhibiting thoughts, disturbing emotions, or memories. EFT regulates the flow of energy in the meridian system of the individual, causing relaxation in the mind, body, and emotions.
Period: Overall Study
Arm/Group | Music Therapy | Emotional Freedom Technique | Control
Started | 32 | 32 | 32
Completed | 30 | 30 | 30
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: This study was conducted with 90 volunteer students studying at the Nursing Department of the Health Sciences Faculty.
Groups:
- Implementation of EFT: The EFT application protocol was explained to the students with the help of the image in the picture for 5 minutes. The method was applied through the investigator tapping on their bodies and the students repeating the steps for three sessions. Each of the treatment sessions was approximately three minutes, resulting in a nine-minute treatment for intervention. Each EFT session was performed by following the steps below.
  The content of each EFT session was as follows:
  1. Preparation
  2. Tapping Series
  3. The Nine Gamut Sequence and Eye Movements
  EFT: EFT includes taps, nine gamut sequences, and eye movements on the meridian system, focusing on the individual's inhibiting thoughts, disturbing emotions, or memories. EFT regulates the flow of energy in the meridian system of the individual, causing relaxation in the mind, body, and emotions.
- Total: Total of all reporting groups
Arm/Group | Implementation of Music Therapy | Implementation of EFT | Control | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.96 (0.88) | 19.1 (0.88) | 19.53 (1.07) | 19.27 (1.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 24 | 74
  Male | 3 | 7 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 30 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Situational-Continuous Anxiety Inventory
Description: The Situational Anxiety Scale was used for scoring anxiety. The Situational-Continuous Anxiety Inventory includes two separate scales with a total of 40 items. This study employed the Situational Anxiety Scale. The Situational Anxiety Scale consists of a total of 20 items. Its reliability coefficient varies between 0.83-0.96. The participants were expected to respond to the items according to their feelings and thoughts at that moment. In this study, the Cronbach's alpha value of the Situational Anxiety Scale was 0.92.
  The items of the Situational Anxiety Scale are scored on a scale of 1-4 depending on the level at which the mentioned emotions or behaviors were experienced. The total score obtained from the scale can vary between 20 and 80. Higher scores indicate higher levels of anxiety.
Time Frame: Immediately after intervention completion, an average of 1 hours
Population: This study was conducted with 90 volunteering students studying at the Faculty of Health Sciences, Department of Nursing, at a foundation university in Medipol University.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Music Therapy | Emotional Freedom Technique | Control
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 44 [41 to 49] | 43 [34 to 51] | 56 [44 to 59]

ADVERSE EVENTS:
Time Frame: 1 day
Description: There was no adverse event during and after interventions.
Groups:
- Music Therapy: For the music therapy, lecturers specializing in music therapy were consulted and accordingly a "mahur maqam," an instrumental piece of traditional Turkish music played on the saz, was chosen. The students listened to this music for about 15 minutes. There was no adverse event during and after the intervention.
- Emotional Freedom Technique (EFT): EFT was applied as follows: first, the researcher tapped on different parts of students' bodies and the students repeated the steps for three sessions. Each of the treatment sessions took approximately three minutes, nine minutes in total. There was no adverse event during and after the intervention.
- Control: For the control group, 15 minutes of free time was given. There was no adverse event during and after the intervention.
Arm/Group | Music Therapy | Emotional Freedom Technique (EFT) | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT03645811/Prot_SAP_000.pdf